CLINICAL TRIAL: NCT02156700
Title: Quantitative Real-time Ultrasound Elastography (Shear Wave Elastography - SWE™) for Characterisation of Liver Tumors
Brief Title: Quantitative Real-time Ultrasound Elastography for Characterisation of Liver Tumors
Status: Completed | Type: Observational
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Ivica Grgurevic, MD, associate professor, University Hospital Dubrava
Other Study IDs: KBD-IG1
Record Dates: First submitted 2014-05-12; First posted 2014-06-05 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Haemangioma; Metastases; Cholangiocellular Carcinoma; Hepatocellular Carcinoma; Focal Nodular Hyperplasia
Keywords: shear wave elastography; haemangiomas; metastases; hepatocellular carcinoma; focal nodular hyperplasia; cholangiocellular carcinoma
MeSH Terms: conditions — Hemangioma, Capillary; Neoplasm Metastasis; Cholangiocarcinoma; Carcinoma, Hepatocellular; Focal Nodular Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver tumors: Measurement of tumor stiffness by Shear wave elastography - SWE™
  Interventions: Procedure: Shear wave elastography

INTERVENTIONS:
Procedure: Shear wave elastography — Measurement of tumor stiffness by Shear wave elastography - SWE™
  Other Names: Shear wave elastography - SWE™

SUMMARY:
Shear Wave Elastography (SWE™) is a quantitative elastography method for measuring tissue stiffness. The difference in stiffness between benign and malignant tumors has been demonstrated by other elastography methods (acoustic radiation force impulse imaging, transient elastography and/or magnetic resonance elastography). The investigators hypothesized that benign liver tumors are softer than malignant liver tumors measured by SWE™, allowing differentiation between the two by tumor stiffness expressed in kilopascal (kPa). In this study benign and malignant liver tumors will be evaluated in five groups: 1) hemangioma and 2) focal nodular hyperplasia (FNH) representing the most common benign liver tumors; 3) metastases and 4) cholangiocarcinoma (CCC), both presenting malignant tumors mostly appearing in otherwise healthy liver, and 5) hepatocellular carcinoma (HCC) mostly occurring in cirrhotic liver, which can potentially influence elastographic measurements therefore querying the appropriateness of comparison between tumors in healthy and cirrhotic liver. Enrolled patients will undergo transabdominal ultrasonography and SWE™ examination. The tumor stiffness will be measured five times for each tumor. Additionally, surrounding liver parenchyma stiffness will be measured. The nature of the liver tumor will be defined through a standard diagnostic workup according to current guidelines, including contrast enhanced multi-slice CT, MRI and/or cytology/histology, as applicable. In the final analysis the mean tumor stiffness and tumor-parenchyma ratio will be calculated for each group as well as for benign and malignant tumors separately, and cut-off values for the differentiation of various groups will be derived. The clinical value of the method will be appraised based on specificity, sensitivity, positive and negative predictive values, and AUC.

ELIGIBILITY:
Inclusion Criteria:

* liver tumors detected on US examination of the liver
* compliance to the study protocol
* signed approval for the diagnostic ultrasound with SWE™

Exclusion Criteria:

* haemangioma, focal nodular hyperplasia (FNH), metastasis, cholangiocellular carcinoma (CCC) or hepatocellular carcinoma (HCC) in the proximity of liver capsule (less than 1 cm from the liver surface)
* haemangioma, FNH, metastasis, CCC or HCC deep in the lever parenchyma (more than 7 cm away from the surface)
* liver tumors other than haemangioma, FNH, metastasis, CCC and HCC
* severe hepatitis defined by alanine aminotransferase (ALT) values > 5 x upper limit of normal (ULN)
* obstructive jaundice
* congestive heart failure
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients and inpatients in a tertiary care hsopital
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Tumor stiffness | at the time of enrollment
  tumor stiffness expressed in kPa, measured by ShearWave ™ Elastography (SWE™) Aixplorer® ultrasound machine from SuperSonic Imagine, Aix-en-Provence, France

SECONDARY OUTCOMES:
tumor to parenchyma stiffness ratio | at the time of enrollment
  comparison between tumor and surrounding liver parenchyma stiffness as expressed by tumor to liver parenchyma stiffness ratio

CONTACTS AND LOCATIONS:
Overall Officials: Ivica Grgurevic, MD, PhD, Principal Investigator — University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

REFERENCES:
- [Background] Masuzaki R, Tateishi R, Yoshida H, Sato T, Ohki T, Goto T, Yoshida H, Sato S, Sugioka Y, Ikeda H, Shiina S, Kawabe T, Omata M. Assessing liver tumor stiffness by transient elastography. Hepatol Int. 2007 Sep;1(3):394-7. doi: 10.1007/s12072-007-9012-7. Epub 2007 Jul 21. PMID 19669335
- [Background] Davies G, Koenen M. Acoustic radiation force impulse elastography in distinguishing hepatic haemangiomata from metastases: preliminary observations. Br J Radiol. 2011 Oct;84(1006):939-43. doi: 10.1259/bjr/97637841. Epub 2011 Mar 8. PMID 21385910
- [Background] Cho SH, Lee JY, Han JK, Choi BI. Acoustic radiation force impulse elastography for the evaluation of focal solid hepatic lesions: preliminary findings. Ultrasound Med Biol. 2010 Feb;36(2):202-8. doi: 10.1016/j.ultrasmedbio.2009.10.009. Epub 2009 Dec 16. PMID 20018432
- [Background] Heide R, Strobel D, Bernatik T, Goertz RS. Characterization of focal liver lesions (FLL) with acoustic radiation force impulse (ARFI) elastometry. Ultraschall Med. 2010 Aug;31(4):405-9. doi: 10.1055/s-0029-1245565. Epub 2010 Jul 22. PMID 20652853